CLINICAL TRIAL: NCT00820807
Title: Novel Fiber Effects on Glucose Metabolism and Insulin Sensitivity for Individuals at High Risk for Diabetes: a Randomized, Placebo-controlled, Double-blind, Parallel Group Clinical Trial
Brief Title: Effects of Novel Fiber on Glucose Homeostasis in Individuals at Risk for Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to a non-safety-related issue with the beverage (test vehicle).
Sponsor: Cargill (Industry)
Responsible Party: Harold E. Bays, MD, FACP/ Medical Director and President, Louisville Metabolic and Atherosclerosis Research Center (LMARC)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CFIS-08-003
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Insulin Resistance
Keywords: dietary fiber; fiber; insulin sensitivity; insulin resistance; glucose metabolism
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 3g/day
  Interventions: Other: Novel dietary fiber
- 2 (Experimental): 6g/day
  Interventions: Other: Novel dietary fiber
- Placebo beverage (Placebo Comparator): 0g/day
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Novel dietary fiber — oral consumption in beverage
  Arms: 1
Other: Novel dietary fiber — oral consumption in beverage
  Arms: 2
Other: Placebo — oral consumption in beverage
  Arms: Placebo beverage

SUMMARY:
This study will critically evaluate the effects of a novel dietary fiber administered to subjects at high risk for developing diabetes to determine if this intervention will improve insulin sensitivity compared to control product administration and, thus, decrease risk for developing diabetes.

The hypothesis is that consuming this novel fiber twice a day for 12 weeks will significantly decrease fasting plasma glucose, insulin and glycosylated hemoglobin values in pre-diabetic subjects (i.e. subjects with fasting plasma glucose levels 95-140 mg/dl at screening) compared to consumption of the control product.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any racial/ethnic group; able to read, comprehend, and write English at a sufficient level to complete study-related materials
* Age: >30 and <65 years at randomization into this trial
* BMI: 25-35 kg/m2 at randomization into this trial
* Fasting blood glucose: 95-140 mg/dl (for those with glucose 95-99mg/dl, must have history of gestational diabetes or first degree relative (parent or sibling) with history of diabetes; for those with glucose 100-125 mg/dl, will be enrolled as the primary target for recruitment; for those with glucose 126-140 mg/dl (asymptomatic diabetes), must not have prior diagnosis of diabetes and must not have prior treatment/pharmacotherapy for diabetes)
* Good general health as evidenced by the medical history
* Blood chemistry and urinalysis results within normal ranges or within an acceptable range determined by the physician on site and/or in consultation with the Medical Monitor
* Available and willing to participate in the study for up to 15 weeks
* Willing to follow a weight-maintaining Lifestyle diet throughout the 12 week trial, maintain physical activity patterns at baseline levels throughout the study period, and not add new exercise routines, dietary supplements, vitamins or other unusual food products
* Willing to consume two 16 oz beverages every day with meals for 12 weeks and able to transport the test article

Exclusion Criteria:

* Presence of any condition the Investigator believes would interfere with subject's ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk
* Food allergy or sensitivity to any of the ingredients in the study product (e.g. Gluten sensitivity, celiac disease)
* Participation in another clinical trial that might interfere with this trial or exposure to any investigational agent within 30 days prior to first visit
* History of diabetes (subjects with a prior history of gestational diabetes may be enrolled if they had no pharmacologic treatment for diabetes since pregnancy)
* Treatment for diabetes or a related condition (e.g., polycystic ovary syndrome) with metformin, an oral agent, or insulin or other injections used for diabetes management
* Uncontrolled hypertension (i.e., systolic blood pressure >160 mm Hg, or a diastolic blood pressure >95 mmHg based on an average of 3 readings sitting)
* Fasting serum triglyceride value >200 mg/dl (since changes in triglyceride values can affect glucose homeostasis)
* Untreated hypothyroidism with a TSH > 1.5 times the upper limit of normal for the test laboratory with repeat value that also exceeds this limit
* Recent history of weight loss (>4 kg in the past 3 months) or a significant variation in weight (>4 kg in the past 3 months, for example, due to a medical condition such as pregnancy, or hormonal therapy)
* Use of medications or herbal remedies for weight loss (e.g., sibutramine, orlistat, amphetamines, phentermine, and ma huang) or use of these substances within the past 3 months
* Current or recent history (past 12 months) of drug, alcohol or chemical abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor)
* Pregnant, breast-feeding or female of child-bearing potential who is unwilling to commit to the use of a medically approved form of contraception throughout the study period.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Mean changes in fasting and post-glucose administration values for plasma glucose from baseline to end of study | 0 weeks, 6 weeks, 9 weeks,12 weeks
Mean changes in fasting and post-glucose administration values for plasma insulin from baseline to end of study | 0 weeks, 6 weeks, 9 weeks,12 weeks
Mean changes in blood HbA1c values from baseline to end of study | 0 weeks, 12 weeks

SECONDARY OUTCOMES:
Mean changes from baseline to end of study in HOMA, a measure of insulin sensitivity | 0 weeks, 6 weeks, 9 weeks,12 weeks
Mean changes from baseline for fasting serum total cholesterol, HDL-cholesterol, LDL-cholesterol and triglyceride values at 6 and 12 weeks | 0 weeks, 6 weeks, 12 weeks
Percentage change and absolute change from baseline in body weight at each treatment visit | 0 weeks, 3 weeks, 6 weeks, 9 weeks, 12 weeks
Mean changes from baseline in waist circumference at selected visits | 0 weeks, 12 weeks
Mean changes in total body fat, lean tissue and abdominal fat as determined by DEXA [distribution or absolute changes] | 0 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harold E Bays, MD, FACP, Principal Investigator — Louisville Metabolic and Atherosclerosis Research Center
Locations (1):
- Louisville Metabolic and Atherosclerosis Research Center (LMARC), Louisville, Kentucky, United States

REFERENCES:
- [Background] Anderson JW, Kendall CW, Jenkins DJ. Importance of weight management in type 2 diabetes: review with meta-analysis of clinical studies. J Am Coll Nutr. 2003 Oct;22(5):331-9. doi: 10.1080/07315724.2003.10719316. PMID 14559925
- [Background] Lindstrom J, Peltonen M, Eriksson JG, Louheranta A, Fogelholm M, Uusitupa M, Tuomilehto J. High-fibre, low-fat diet predicts long-term weight loss and decreased type 2 diabetes risk: the Finnish Diabetes Prevention Study. Diabetologia. 2006 May;49(5):912-20. doi: 10.1007/s00125-006-0198-3. Epub 2006 Mar 16. PMID 16541277
- [Background] Weickert MO, Mohlig M, Schofl C, Arafat AM, Otto B, Viehoff H, Koebnick C, Kohl A, Spranger J, Pfeiffer AF. Cereal fiber improves whole-body insulin sensitivity in overweight and obese women. Diabetes Care. 2006 Apr;29(4):775-80. doi: 10.2337/diacare.29.04.06.dc05-2374. PMID 16567814
- [Background] Murtaugh MA, Jacobs DR Jr, Jacob B, Steffen LM, Marquart L. Epidemiological support for the protection of whole grains against diabetes. Proc Nutr Soc. 2003 Feb;62(1):143-9. doi: 10.1079/pns2002223. PMID 12740069
- [Background] Anderson JW, Conley SB, Nicholas AS. One hundred pound weight losses with an intensive behavioral program: changes in risk factors in 118 patients with long-term follow-up. Am J Clin Nutr. 2007 Aug;86(2):301-7. doi: 10.1093/ajcn/86.2.301. PMID 17684198
- [Background] Lu ZX, Walker KZ, Muir JG, Mascara T, O'Dea K. Arabinoxylan fiber, a byproduct of wheat flour processing, reduces the postprandial glucose response in normoglycemic subjects. Am J Clin Nutr. 2000 May;71(5):1123-8. doi: 10.1093/ajcn/71.5.1123. PMID 10799374
- [Background] Behall KM, Scholfield DJ, Hallfrisch J. Comparison of hormone and glucose responses of overweight women to barley and oats. J Am Coll Nutr. 2005 Jun;24(3):182-8. doi: 10.1080/07315724.2005.10719464. PMID 15930484
- [Background] Jenkins AL, Jenkins DJ, Zdravkovic U, Wursch P, Vuksan V. Depression of the glycemic index by high levels of beta-glucan fiber in two functional foods tested in type 2 diabetes. Eur J Clin Nutr. 2002 Jul;56(7):622-8. doi: 10.1038/sj.ejcn.1601367. PMID 12080401
- [Background] Vuksan V, Sievenpiper JL, Owen R, Swilley JA, Spadafora P, Jenkins DJ, Vidgen E, Brighenti F, Josse RG, Leiter LA, Xu Z, Novokmet R. Beneficial effects of viscous dietary fiber from Konjac-mannan in subjects with the insulin resistance syndrome: results of a controlled metabolic trial. Diabetes Care. 2000 Jan;23(1):9-14. doi: 10.2337/diacare.23.1.9. PMID 10857960
- [Background] Kim JI, Kim JC, Kang MJ, Lee MS, Kim JJ, Cha IJ. Effects of pinitol isolated from soybeans on glycaemic control and cardiovascular risk factors in Korean patients with type II diabetes mellitus: a randomized controlled study. Eur J Clin Nutr. 2005 Mar;59(3):456-8. doi: 10.1038/sj.ejcn.1602081. PMID 15536472
- [Background] Vuksan V, Jenkins DJ, Spadafora P, Sievenpiper JL, Owen R, Vidgen E, Brighenti F, Josse R, Leiter LA, Bruce-Thompson C. Konjac-mannan (glucomannan) improves glycemia and other associated risk factors for coronary heart disease in type 2 diabetes. A randomized controlled metabolic trial. Diabetes Care. 1999 Jun;22(6):913-9. doi: 10.2337/diacare.22.6.913. PMID 10372241
- [Background] American Heart Association Nutrition Committee; Lichtenstein AH, Appel LJ, Brands M, Carnethon M, Daniels S, Franch HA, Franklin B, Kris-Etherton P, Harris WS, Howard B, Karanja N, Lefevre M, Rudel L, Sacks F, Van Horn L, Winston M, Wylie-Rosett J. Diet and lifestyle recommendations revision 2006: a scientific statement from the American Heart Association Nutrition Committee. Circulation. 2006 Jul 4;114(1):82-96. doi: 10.1161/CIRCULATIONAHA.106.176158. Epub 2006 Jun 19. PMID 16785338
- [Background] Keenan JM, Goulson M, Shamliyan T, Knutson N, Kolberg L, Curry L. The effects of concentrated barley beta-glucan on blood lipids in a population of hypercholesterolaemic men and women. Br J Nutr. 2007 Jun;97(6):1162-8. doi: 10.1017/S0007114507682968. Epub 2007 Apr 20. PMID 17445284